CLINICAL TRIAL: NCT03716414
Title: Evaluation of the Efficacy for Sentinel Lymph Node Policy in High-risk Endometrial Carcinoma
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Principal Investigator, Fudan University
Other Study IDs: 53201016
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Endometrial Adenocarcinoma
Keywords: Sentinel lymph node

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental SLN arm: Experimental SLN arm
  1. Intra-operative sentinel lymph node (SLN) mapping with indocyanine green injected into the stroma of the cervix.
  2. Full bilateral laparoscopic lymphadenectomy and hysterectomy:
  If bilateral SLN are detected, all positive SLN will be removed. Then the surgeons proceed to a total hysterectomy, bilateral salpingo-oophorectomy, and lymphadenectomy including complete pelvic lymphadenectomy and aortic lymph node dissection.
  If only unilateral SLN or non SLN are detected, surgeons will proceed to complete pelvic lymphadenectomy and aortic lymph node dissection.
  Interventions: Procedure: SLN mapping

INTERVENTIONS:
Procedure: SLN mapping — Intra-operative SLN mapping with indocyanine green: Intracervical injection will be performed by the surgeon. Sub-mucous injections will be performed with 50% diluted dye at 3 and 9 o'clock positions. 1ml injection contained infracyanine green will be injected deeply into the stroma of the cervix (1cm-depth), and Arms Assigned Interventions another 1ml will be injected superficially (2mm-depth).
  The time between the injection and the search for SLN must be as soon as possible.

SUMMARY:
To evaluate the efficacy of sentinel lymph node biopsy technique in patients with high-risk endometrial carcinoma, which provides the evidence that sentinel lymph node biopsy technique could substitute the systematic Lymph node dissection(LND).

DETAILED DESCRIPTION:
Comprehensive surgical staging for endometrial carcinoma(EC) is an indisputable staging and prognostic tool. The staging procedure includes total hysterectomy, bilateral salpingo-oophorectomy, and lymphadenectomy, omental biopsy if necessary. Since lymph node metastasis is one of the most important risk factors of prognosis. The dissection of lymph nodes has been used for staging, prognostic information, and to determine the need for adjuvant therapy. The approach to lymph node evaluation in women with EC is still a subject of debate. Practice varies across different institutions or surgeons. In general, the options for management of retroperitoneal lymph nodes include no lymph node dissection (LND), systematic LND only if the risk of lymph node metastasis exceeds a certain threshold, or routine sentinel LND following lymphatic mapping. lymphadenectomy is significantly associated with longer operating time, higher surgical costs, greater rate of infection, as well as the occurrence of lymphocysts and lymphedema, moreover, there is lack of evidence of a therapeutic benefit of LND, less invasive techniques have emerged as possible alternatives. The technique for lymphatic mapping and sentinel lymph node dissection (SLND) in EC has been refined and found a low false-negative rate for detection of positive lymph nodes. The 2018 National Comprehensive cancer Network (NCCN) guideline of uterus cancer states SLN mapping can be considered for the surgical staging of apparent uterine-confined malignancy when there is no metastasis demonstrated by imaging studies or no obvious extrauterine disease at exploration. It indicates low-risk patients could avoid those side effects of the systematic Lymph node dissection. Whether high-risk patients (grade 3, deep myometrial invasion, non-endometrioid endometrial cancer, and Cervical invasion) can be benefited from this technique? This prospective cohort study is designed to To evaluate the efficacy of sentinel lymph node biopsy technique in patients with high-risk endometrial carcinoma. Surgery should be performed within a maximum of 4 weeks from the patient's first consultation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~100 years.
2. No contraindication to surgery.
3. Signed and dated informed consent.
4. high-risk endometrial cancer with grade 3, deep myometrial invasion, non-endometrioid endometrial cancer, and Cervical invasion (in intraoperative frozen section examinations).
5. With any suspicious pelvic, para-aortic or distant lymph node metastasis in preoperative imaging tests including MRI/CT/positron emission computed tomography(PET)-CT.

Exclusion Criteria:

1. Low-risk endometrioid endometrial cancer with grade 1-2, superficial myometrial invasion and tumor diameter < 2cm (in intraoperative frozen section examinations).
2. Intermediate-risk endometrioid endometrial cancer with grade 1-2, superficial myometrial invasion and tumor diameter ≥ 2cm (in intraoperative frozen section examinations).

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-100 years old with high-risk endometrial carcinoma (grade 3 endometroid endometrial cancer, deep myometrial invasion, non-endometrioid endometrial cancer, and Cervical invasion (in intraoperative frozen section examinations) and without no contraindication to surgery will be recruited.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-16 (Actual)

PRIMARY OUTCOMES:
Performance Analysis | Within 14 days after the surgery
  Using the final pathological diagnosis as the Gold Standard, the investigators will calculate the sensitivity, specificity, and predictive accuracy of mapping and detection of SLN with metastatic disease.

SECONDARY OUTCOMES:
Postoperative complications | 1 years after the surgery
  calculate the incidence of complications such as lymph cysts, lymph edema, and postoperative fever etc.
Recurrence rate | 5 years after the surgery
  The recurrence rate will be followed up.
Adjuvant therapy rate | 5 years after the surgery
  The adjuvant therapy rate will be followed up.
5-year survival rate | 5 years after the surgery
  The 5-year survival rate will be followed up.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Wang, Ph.D., Study Director — Obstetrics and Gynecology Hospital, Fudan University; Xuezhen Luo, Ph.D., Principal Investigator — Obstetrics and Gynecology Hospital, Fudan University; Xiaojun Chen, Ph.D., Study Chair — Obstetrics and Gynecology Hospital, Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided